CLINICAL TRIAL: NCT02560740
Title: A Randomised, Double-blinded, Placebo Controlled Study to Assess the Efficacy and Safety of PerOx Quench or Placebo for 35 Days on the Prevention of Oxaliplatin Treatment Induced Sensory Neuropathy
Brief Title: A Study of the Efficacy and Safety of PerOx Quench on the Prevention of Oxaliplatin Treatment Induced Neuropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subjects' not-well compliance due to diarrhea and softening stool after taking PerOx Quench 4 sachets a day.
Sponsor: SMR Biotech Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POQ 00001
Record Dates: First submitted 2015-08-15; First posted 2015-09-25 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer; Advanced Gastric Cancer; Neuropathy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PerOx Arm (Experimental): PerOx Quench arm 4g/sachet each time by water, q6h
  Interventions: Dietary Supplement: PerOx Quench
- Comparative Arm (Placebo Comparator): PerOx Quench placebo 4g/sachet each time by water, q6h
  Interventions: Dietary Supplement: PerOx Quench Placebo

INTERVENTIONS:
Dietary Supplement: PerOx Quench — By 1 week pretreatment of PerOx Quench and following 4 weeks taken to decrease the CIPN incidence.
  Arms: PerOx Arm
Dietary Supplement: PerOx Quench Placebo — By 1 week pretreatment of Placebo and following 4 weeks taken to record the CIPN incidence.
  Arms: Comparative Arm

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a progressive, enduring, and often irreversible condition featuring pain, numbness, tingling and sensitivity to cold in the hands and feet (sometimes progressing to the arms and legs) that afflicts between 30 and 40 percent of patients undergoing chemotherapy.

American Society of Clinical Oncology (ASCO) guidance on The Journal of Clinical Oncology (JCO, 2014 April 14) does not recommend any prophylaxis regimen for CIPN.

PerOx Quench has unique membrane protection and anti-oxidative function as a special food, that's why to try to explore its preventive effects on CIPN prevention induced by Oxaliplatin for colorectal cancer or gastric cancer chemotherapy.

DETAILED DESCRIPTION:
This study uses two stage group-sequential sampling design, based on current data, assumed the CIPN incidence rate is 50% in placebo arm, while 20% in PerOx Quench arm（60% reduction）, set a=0.05，80％ power, random allocation ratio is 1:1, obtained the subjects number is 41（total 82) by PASS 11 software for superior design; considering 10% drop out rate, final number of subjects totally is 90.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80 years old, male and female
2. Without anti-cancer treatment before randomization, ECOG score 0-2
3. Estimate to bear at least 4 cycles chemotherapy treatment with normal function of heart, lungs, liver and kidneys.
4. Survival expectation ≥6 months
5. Signed Informed Consent Form, willing to follow all study procedures

Exclusion Criteria:

1. Received chemotherapy treatment within 4 weeks before randomization.
2. Current peripheral neuropathy(by chemotherapy, diabetes mellitus, alcoholic disease) and relative symptoms with relevant treatment.
3. Concurrent treatment within 30 days after randomization with the following drugs: Calcium-Magnesium injection, glutathione, and similar ingredients with PerOx Quench (such as polyene phosphatidyl choline).
4. Laboratory tests found not suitable for chemotherapy patients (Absolute neutrophil count <2.0×10*9/L<2,000/mm3>; or platelet count<100× 10*9/L<100,000/mm3>; or hemoglobin <10/dl; or serum total bilirubin >2 Upper Limit Of Normal (ULN), alanine aminotransferase (ALT)/aspartate aminotransferase (AST)>3 Upper Limit Of Normal (ULN); or serum creatinine >1.5 Upper Limit Of Normal (ULN) <or creatinine clearance rate

   ≤60ml/min>）.
5. Pregnancy, lactation and reluctant to using contraception women.
6. Patients with symptomatic brain metastases and other mental disorders could not be self assessment.
7. Alcohol and/or drug abuse or doctors determine compliance's claim.
8. Within a month in other clinical trial subjects.
9. Once into the group of this study, or random within eight weeks before using this product.
10. personnel involved this study.
11. Not completed independent self assessment of patients.
12. Other researchers determine does not fit to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of Oxaliplatin-induced Peripheral Neuropathy incidence rate on the 35 day in 2 arms. | 35 day after randomization
  Peripheral neuropathy incidence rate was measured by frequency and percentage of any Oxaliplatin-induced Peripheral Neuropathy symptoms.

SECONDARY OUTCOMES:
Evaluation of Oxaliplatin-induced Peripheral Neuropathy severity by PI on the 35 day in 2 arms. | 35 day after randomization
  Peripheral neuropathy severity by PI was measured by each related symptom grading, and the most serious symptom will be evaluated by National Cancer Institute Common Toxicity Criteria (NCI-CTC) classification.
Evaluation of Oxaliplatin-induced Peripheral Neuropathy severity by subjects on the 35 day in 2 arms. | 35 day after randomization
  Peripheral neuropathy severity by subjects was measured by Visual Analogue Scale (VAS) score (Scores range from 0 [no symptom] to 10 [worst possible symptom]).
Evaluation of subjects quality of life difference in 2 arms on the 35 day. | 35 day after randomization
  Quality of Life (QoL) will be measured by European Organization for Research and Treatment of Cancer quality of life questionaire C30 (EORTCQLQ-C30) questionnaire.
Evaluation of subjects Eastern Cooperation Oncology Group-Performance Score (ECOG-PS) difference in 2 arms on the 35 day. | 35 day after randomization
  Eastern Cooperation Oncology Group-Performance Score (ECOG-PS) will be measured by ECOG-PS score.
Evaluation of the Adverse Events (AEs) incidence rate on 35 day in 2 arms. | Sign ICF to 35 day after randomization
  The Adverse Events (AEs) incidence rate was measured by frequency and percentage of participants with Treatment-Related Grade 3 or above Adverse Events during this trial. The grade of Adverse Events was assessed by Common Toxicity Criteria Adverse Event (CTCAE) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jiejun WANG, MD., Ph.D, Study Director — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No